CLINICAL TRIAL: NCT01446224
Title: Postmarketing Cardiovascular Ischemia and Torsades de Pointes Monitoring for Pazopanib Using Observational Databases
Brief Title: Cardiovascular and Torsades de Pointes Monitoring for Pazopanib
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 114428; WEUKSTV4602 (Other: GSK)
Record Dates: First submitted 2011-10-03; First posted 2011-10-05 (Estimated); Last update posted 2015-03-27 (Estimated); Status verified 2015-03

CONDITIONS: Carcinoma, Renal Cell
Keywords: adverse events; pazopanib; Torsades des Pointes; renal cell carcinoma; anti-VEGF agents; observational data; cardiac ischemia
MeSH Terms: conditions — Carcinoma, Renal Cell; Coronary Artery Disease | interventions — pazopanib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Subjects who experience cardiac ischemia: Subjects who experience cardiac ischemia including myocardial infarction, unstable angina, transient ischemic attack, and cerebrovascular accident
  Interventions: Drug: Pazopanib; Drug: Other anti-VEGFs
- Subjects who do not experience cardiac ischemia: Subjects who do not experience cardiac ischemia
  Interventions: Drug: Pazopanib; Drug: Other anti-VEGFs
- Subjects who experience Torsades de Pointes: Subjects who experience Torsades de Pointes
  Interventions: Drug: Pazopanib; Drug: Other anti-VEGFs
- Subjects who do not experience Torsades de Pointes: Subjects who do not experience Torsades de Pointes
  Interventions: Drug: Pazopanib; Drug: Other anti-VEGFs

INTERVENTIONS:
Drug: Pazopanib — Patients treated with pazopanib
Drug: Other anti-VEGFs — Patients treated with other anti-VEGFs including Bevacizumab, Sorafenib, and Sunitinib

SUMMARY:
This observational study is conducted as part of a systematic pharmacovigilance activity, to provide a population-based context for Pazopanib use outside of the clinical trial setting. The aims of the study are to examine the incidence of cardiovascular ischemia (including myocardial infarction, unstable angina, transient ischemic attack, and cerebrovascular accident) and cardiac arrhythmia (Torsades de Pointes) in renal cell carcinoma patients treated with marketed anti-VEGF agents [Pazopanib (VOTRIENT), Bevacizumab (AVASTIN), Sorafenib (NEXAVAR), and Sunitinib (SUTENT)].

Two databases will be utilized for this study: a large healthcare claims database in the U.S. and the Dutch linked medical registries (PHARMO RLS). The databases will provide large, geographically varied, non-trial populations in which to examine the incidence of the stated cardiovascular ischemic events and Torsades des Pointes.

ELIGIBILITY:
Inclusion Criteria:

The anti-VEGF cohorts will include patients with the following characteristics:

* Adult patients (age ≥18 years)
* Prescribed or administered an anti-VEGF agent: Pazopanib, Bevacizumab, Sorafenib or Sunitinib on or after approval date of Pazopanib
* Diagnosed with renal cell cancer

Exclusion Criteria:

* Patients with multiple primary cancer diagnoses

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study cohorts will be created in two healthcare databases to follow the outcomes of interest in (i) Pazopanib users, and (ii) users of other marketed anti-VEGF drugs (Bevacizumab, Sorafenib, Sunitinib).
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2010-12; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Cardiovascular ischemia | Over four years from approval of pazopanib
  Cardiovascular ischemia including myocardial infarction, unstable angina, transient ischemic attack, and cerebrovascular accident

SECONDARY OUTCOMES:
Torsades de Pointes | Over four years from approval of pazopanib
  Torsades de Pointes

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline